CLINICAL TRIAL: NCT00234884
Title: A Five-year, Post-marketing Observational Study to Follow-up Patients With Rheumatoid Arthritis Formerly Treated in Study M02-497 (ReAct) and Subsequently Prescribed Humira
Brief Title: Post-marketing Observational Study in Subjects With Rheumatoid Arthritis
Acronym: ReAlise
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: M03-634
Record Dates: First submitted 2005-09-16; First posted 2005-10-10 (Estimated); Results first posted 2011-09-30 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adalimumab: RA patients in treatment with commercial adalimumab
  Interventions: Biological: adalimumab

INTERVENTIONS:
Biological: adalimumab — commercial adalimumab as prescribed by the rheumatologist in a normal clinical setting and in accordance with the Summary of Product Characteristics (SmPC)
  Other Names: HUMIRA®

SUMMARY:
The purpose of this observational study was to observe and assess the long term use, safety, and effectiveness of adalimumab in a normal clinical setting.

DETAILED DESCRIPTION:
This was a multicenter, uncontrolled, 5-year observational study of adalimumab in the treatment of patients with rheumatoid arthritis (RA) who had received adalimumab for at least 3 months in NCT00448383 (Study M02-497), an interventional study that ended when adalimumab became commercially available for the treatment of RA. Participants had to have been receiving ongoing adalimumab treatment at the time NCT00448383 (Study M02-497) ended and been prescribed commercial adalimumab, and could have received commercial adalimumab for up to 1 year afterward prior to enrollment in NCT00234884 (Study M03-634).

Physician investigators were encouraged to treat participants as they would any other patient with RA in their routine clinical practice, and were free to determine the appropriate therapy for each patient. Concomitant treatment with disease-modifying antirheumatic drugs (DMARDs), including methotrexate, could be continued while receiving adalimumab. If treatment with adalimumab was permanently discontinued for any reason, participants were discontinued from the study and the reason was recorded. Investigators were asked to record adverse events up to 3 months after last administration of adalimumab.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ongoing adalimumab treatment who completed at least Month 3 (Visit 5) of NCT00448383 (Study M02-497) and who had subsequently been prescribed adalimumab according to the Summary of Product Characteristics (SmPC).
* Participants must have been willing to consent to data being collected and provided to Abbott.

Exclusion Criteria:

· Participants with contraindications according to the SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were patients with rheumatoid arthritis (RA) who had received adalimumab for at least 3 months in NCT00448383 (Study M02-497) and had been prescribed commercial adalimumab following termination of that study. At the time of enrollment in NCT00448383 (Study M02-497), participants had failed one or more disease-modifying antirheumatic drugs (DMARDs) and had active, moderate to severe RA despite concurrent RA treatment.
Sampling Method: Non-Probability Sample
Enrollment: 3435 (Actual)
Dates: Start 2003-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, PhD, Study Director — Abbott
Locations (311):
- Australia (6):
  - Site Ref # / Investigator 5606, Camperdown, New South Wales
  - Site Ref # / Investigator 49504, New Lambton, New South Wales
  - Site Ref # / Investigator 49508, Brisbane, Queensland
  - Site Ref # / Investigator 49505, Woodville, South Australia
  - Site Ref # / Investigator 49503, West Heidelberg, Victoria
  - Site Ref # / Investigator 49502, Cairns
- Austria (12):
  - Site Ref # / Investigator 49747, Bad Schallerbach
  - Site Ref # / Investigator 49517, Graz
  - Site Ref # / Investigator 49521, Graz
  - Site Ref # / Investigator 49518, Innsbruck
  - Site Ref # / Investigator 49746, Klagenfurt
  - Site Ref # / Investigator 49748, Laab im Walde
  - Site Ref # / Investigator 49516, Linz
  - Site Ref # / Investigator 49523, Oberpullendorf
  - Site Ref # / Investigator 49745, Sankt Pölten
  - Site Ref # / Investigator 49519, Stockerau
  - Site Ref # / Investigator 49520, Vienna
  - Site Ref # / Investigator 4961, Vienna
- Belgium (45):
  - Site Ref # / Investigator 49794, Aalst
  - Site Ref # / Investigator 49817, Antwerp
  - Site Ref # / Investigator 49788, Assebroek
  - Site Ref # / Investigator 49764, Baudour
  - Site Ref # / Investigator 49808, Belsele
  - Site Ref # / Investigator 49806, Bonheiden
  - Site Ref # / Investigator 49809, Bonheiden
  - Site Ref # / Investigator 49798, Braine-l'Alleud
  - Site Ref # / Investigator 49773, Bruges
  - Site Ref # / Investigator 49774, Brussels
  - Site Ref # / Investigator 49763, Brussels
  - Site Ref # / Investigator 49791, Brussels
  - Site Ref # / Investigator 49762, Brussels
  - Site Ref # / Investigator 49811, Brussels
  - Site Ref # / Investigator 49807, Brussels
  - Site Ref # / Investigator 49772, Brussels
  - Site Ref # / Investigator 49780, Chimay
  - Site Ref # / Investigator 49795, Destelbergen
  - Site Ref # / Investigator 49768, Edegem
  - Site Ref # / Investigator 49776, Genk
  - Site Ref # / Investigator 49813, Genk
  - Site Ref # / Investigator 26424, Ghent
  - Site Ref # / Investigator 49766, Gosselies
  - Site Ref # / Investigator 49781, Hamme
  - Site Ref # / Investigator 49814, Hasselt
  - Site Ref # / Investigator 49810, Hasselt
  - Site Ref # / Investigator 49777, Kortrijk
  - Site Ref # / Investigator 49767, La Louvière
  - Site Ref # / Investigator 49801, La Louvière
  - Site Ref # / Investigator 49816, Leuven
  - Site Ref # / Investigator 49775, Lier
  - Site Ref # / Investigator 49789, Liège
  - Site Ref # / Investigator 49778, Lokeren
  - Site Ref # / Investigator 49771, Mechelen
  - Site Ref # / Investigator 49815, Mechelen
  - Site Ref # / Investigator 49796, Merksem
  - Site Ref # / Investigator 49785, Mons
  - Site Ref # / Investigator 49891, Montignies-sur-Sambre
  - Site Ref # / Investigator 49770, Namur
  - Site Ref # / Investigator 49783, Namur
  - Site Ref # / Investigator 49797, Nukerke
  - Site Ref # / Investigator 49787, Ostend
  - Site Ref # / Investigator 49802, Ottignies
  - Site Ref # / Investigator 49793, Sijsele
  - Site Ref # / Investigator 49805, Sint-Niklaas
- France (81):
  - Site Ref # / Investigator 49615, Aix-en-Provence
  - Site Ref # / Investigator 49332, Aix-les-Bains
  - Site Ref # / Investigator 49350, Angers
  - Site Ref # / Investigator 49604, Aulnay-sous-Bois
  - Site Ref # / Investigator 49340, Belfort
  - Site Ref # / Investigator 49621, Berck
  - Site Ref # / Investigator 49339, Besançon
  - Site Ref # / Investigator 49351, Bobigny
  - Site Ref # / Investigator 49365, Bordeaux
  - Site Ref # / Investigator 49611, Boulogne-Billancourt
  - Site Ref # / Investigator 49622, Bourg-en-Bresse
  - Site Ref # / Investigator 49329, Brest
  - Site Ref # / Investigator 49334, Caen
  - Site Ref # / Investigator 49358, Cahors
  - Site Ref # / Investigator 49607, Cannes
  - Site Ref # / Investigator 49612, Carcassonne
  - Site Ref # / Investigator 49628, Cherbourg
  - Site Ref # / Investigator 49613, Clermont-Ferrand
  - Site Ref # / Investigator 49624, Colombes
  - Site Ref # / Investigator 49376, Compiègne
  - Site Ref # / Investigator 49356, Corbeil-Essonnes
  - Site Ref # / Investigator 49370, Créteil
  - Site Ref # / Investigator 49605, Dijon
  - Site Ref # / Investigator 49608, Gleizé
  - Site Ref # / Investigator 49610, Gonesse
  - Site Ref # / Investigator 49379, Grenoble
  - Site Ref # / Investigator 49361, Grenoble
  - Site Ref # / Investigator 49614, La Roche-sur-Yon
  - Site Ref # / Investigator 49601, La Rochelle
  - Site Ref # / Investigator 49373, Le Kremlin-Bicêtre
  - Site Ref # / Investigator 49375, Le Mans
  - Site Ref # / Investigator 49325, Libourne
  - Site Ref # / Investigator 49620, Liévin
  - Site Ref # / Investigator 49360, Lille
  - Site Ref # / Investigator 49623, Limoges
  - Site Ref # / Investigator 49333, Lomme
  - Site Ref # / Investigator 49355, Lunel
  - Site Ref # / Investigator 49337, Lyon
  - Site Ref # / Investigator 49363, Lyon
  - Site Ref # / Investigator 49364, Lyon
  - Site Ref # / Investigator 49603, Mantes-la-Jolie
  - Site Ref # / Investigator 49626, Marseille
  - Site Ref # / Investigator 49342, Marseille
  - Site Ref # / Investigator 49345, Marseille
  - Site Ref # / Investigator 49362, Marseille
  - Site Ref # / Investigator 49330, Montivilliers
  - Site Ref # / Investigator 49323, Montpellier
  - Site Ref # / Investigator 5590, Mulhouse
  - Site Ref # / Investigator 49374, Nantes
  - Site Ref # / Investigator 49642, Narbonne
  - Site Ref # / Investigator 49353, Nice
  - Site Ref # / Investigator 49618, Orange
  - Site Ref # / Investigator 49331, Orléans
  - Site Ref # / Investigator 49326, Paris
  - Site Ref # / Investigator 49600, Paris
  - Site Ref # / Investigator 49625, Paris
  - Site Ref # / Investigator 49359, Paris
  - Site Ref # / Investigator 49352, Paris
  - Site Ref # / Investigator 49343, Pau
  - Site Ref # / Investigator 49344, Pessac
  - Site Ref # / Investigator 49606, Pierre-Bénite
  - Site Ref # / Investigator 49602, Poissy
  - Site Ref # / Investigator 49349, Poitiers
  - Site Ref # / Investigator 49627, Provins
  - Site Ref # / Investigator 49382, Reims
  - Site Ref # / Investigator 49328, Rennes
  - Site Ref # / Investigator 49619, Roubaix
  - Site Ref # / Investigator 49372, Rouen
  - Site Ref # / Investigator 49609, Saint-Aubin-lès-Elbeuf
  - Site Ref # / Investigator 49327, Saint-Brieuc
  - Site Ref # / Investigator 49598, Saint-Etienne
  - Site Ref # / Investigator 49336, Saint-Maurice
  - Site Ref # / Investigator 49346, Strasbourg
  - Site Ref # / Investigator 49366, Thionville
  - Site Ref # / Investigator 49616, Toulon
  - Site Ref # / Investigator 49322, Toulouse
  - Site Ref # / Investigator 49348, Toulouse
  - Site Ref # / Investigator 49324, Tours
  - Site Ref # / Investigator 49617, Valence
  - Site Ref # / Investigator 49371, Valenciennes
  - Site Ref # / Investigator 49629, Vannes
- Germany (48):
  - Site Ref # / Investigator 49573, Aachen
  - Site Ref # / Investigator 49454, Berlin
  - Site Ref # / Investigator 49705, Berlin
  - Site Ref # / Investigator 49480, Berlin
  - Site Ref # / Investigator 49433, Berlin
  - Site Ref # / Investigator 49577, Bremen
  - Site Ref # / Investigator 49451, Chemnitz
  - Site Ref # / Investigator 49551, Cologne
  - Site Ref # / Investigator 5602, Cottbus
  - Site Ref # / Investigator 49441, Damp
  - Site Ref # / Investigator 49446, Dresden
  - Site Ref # / Investigator 49474, Dresden
  - Site Ref # / Investigator 49483, Duisburg
  - Site Ref # / Investigator 49455, Erfurt
  - Site Ref # / Investigator 49579, Erlangen
  - Site Ref # / Investigator 49475, Erlangen
  - Site Ref # / Investigator 49481, Essen
  - Site Ref # / Investigator 49469, Freiburg im Breisgau
  - Site Ref # / Investigator 49711, Freiburg im Breisgau
  - Site Ref # / Investigator 49556, Fürth
  - Site Ref # / Investigator 49482, Gyhum
  - Site Ref # / Investigator 49422, Halle
  - Site Ref # / Investigator 49468, Hamburg
  - Site Ref # / Investigator 49552, Hamburg
  - Site Ref # / Investigator 49466, Hattingen
  - Site Ref # / Investigator 49544, Herrsching am Ammersee
  - Site Ref # / Investigator 49548, Hildesheim
  - Site Ref # / Investigator 49587, Hofheim
  - Site Ref # / Investigator 49447, Jena
  - Site Ref # / Investigator 49431, Leipzig
  - Site Ref # / Investigator 49424, Ludwigsburg
  - Site Ref # / Investigator 49557, Ludwigshafen
  - Site Ref # / Investigator 49704, Marl
  - Site Ref # / Investigator 49547, Mönchengladbach
  - Site Ref # / Investigator 49450, Munich
  - Site Ref # / Investigator 49563, Munich
  - Site Ref # / Investigator 49440, Münster
  - Site Ref # / Investigator 49442, Passau
  - Site Ref # / Investigator 49549, Ratingen
  - Site Ref # / Investigator 49708, Rostock
  - Site Ref # / Investigator 49558, Schlangenbad
  - Site Ref # / Investigator 49445, Sendenhorst
  - Site Ref # / Investigator 49437, Stuttgart
  - Site Ref # / Investigator 49560, Tübingen
  - Site Ref # / Investigator 49460, Villingen
  - Site Ref # / Investigator 49456, Vogelsang-Gommern
  - Site Ref # / Investigator 49449, Wuppertal
  - Site Ref # / Investigator 49545, Würzburg
- Greece (15):
  - Site Ref # / Investigator 49580, Athens
  - Site Ref # / Investigator 49568, Athens
  - Site Ref # / Investigator 49584, Athens
  - Site Ref # / Investigator 49554, Athens
  - Site Ref # / Investigator 49565, Athens
  - Site Ref # / Investigator 49583, Athens
  - Site Ref # / Investigator 49585, Athens
  - Site Ref # / Investigator 49564, Heraklion
  - Site Ref # / Investigator 49567, Ioannina
  - Site Ref # / Investigator 49581, Larissa
  - Site Ref # / Investigator 26425, Pátrai
  - Site Ref # / Investigator 49566, Thessaloniki
  - Site Ref # / Investigator 49582, Thessaloniki
  - Site Ref # / Investigator 49553, Thessaloniki
  - Site Ref # / Investigator 49569, Thessaloniki
- Italy (39):
  - Site Ref # / Investigator 49990, Acqui Terme (AL)
  - Site Ref # / Investigator 49591, Arenzano (GE)
  - Site Ref # / Investigator 49983, Bari
  - Site Ref # / Investigator 49593, Bologna
  - Site Ref # / Investigator 49980, Brescia
  - Site Ref # / Investigator 49986, Cagliari
  - Site Ref # / Investigator 50056, Ferrara
  - Site Ref # / Investigator 49987, Florence
  - Site Ref # / Investigator 49597, Foggia
  - Site Ref # / Investigator 49824, Genoa
  - Site Ref # / Investigator 50051, Genoa
  - Site Ref # / Investigator 49981, Jesi (Ancona)
  - Site Ref # / Investigator 49588, Messina
  - Site Ref # / Investigator 49976, Milan
  - Site Ref # / Investigator 50052, Milan
  - Site Ref # / Investigator 49596, Milan
  - Site Ref # / Investigator 49985, Modena
  - Site Ref # / Investigator 49949, Naples
  - Site Ref # / Investigator 49595, Novara
  - Site Ref # / Investigator 49947, Padua
  - Site Ref # / Investigator 49948, Palermo
  - Site Ref # / Investigator 49978, Perugia
  - Site Ref # / Investigator 49974, Pescara
  - Site Ref # / Investigator 49592, Pisa
  - Site Ref # / Investigator 49992, Potenza
  - Site Ref # / Investigator 49822, Prato
  - Site Ref # / Investigator 49946, Reggio Emilia
  - Site Ref # / Investigator 49989, Rome
  - Site Ref # / Investigator 49950, Rome
  - Site Ref # / Investigator 50057, Rome
  - Site Ref # / Investigator 49984, Rozzano
  - Site Ref # / Investigator 49991, San Cesario Lecce
  - Site Ref # / Investigator 49994, Torino
  - Site Ref # / Investigator 49825, Udine
  - Site Ref # / Investigator 26422, Valeggio Sul Mincio Verona
  - Site Ref # / Investigator 49594, Varese
  - Site Ref # / Investigator 50055, Verbania Pallanza
  - Site Ref # / Investigator 49589, Verona
  - Site Ref # / Investigator 50053, Vimercate
- Netherlands (16):
  - Site Ref # / Investigator 49904, Alkmaar
  - Site Ref # / Investigator 49909, Almere Stad
  - Site Ref # / Investigator 49831, Amersfoort
  - Site Ref # / Investigator 49906, Bergen op Zoom
  - Site Ref # / Investigator 49907, Breda
  - Site Ref # / Investigator 49910, Den Helder
  - Site Ref # / Investigator 49835, Flushing
  - Site Ref # / Investigator 49902, Goes
  - Site Ref # / Investigator 49829, Leeuwarden
  - Site Ref # / Investigator 26426, Rotterdam
  - Site Ref # / Investigator 49830, Rotterdam
  - Site Ref # / Investigator 49908, Schiedam
  - Site Ref # / Investigator 49905, The Hague
  - Site Ref # / Investigator 49920, The Hague
  - Site Ref # / Investigator 49827, Utrecht
  - Site Ref # / Investigator 49903, Venlo
- Portugal (7):
  - Site Ref # / Investigator 49514, Coimbra
  - Site Ref # / Investigator 49515, Lisbon
  - Site Ref # / Investigator 49509, Lisbon
  - Site Ref # / Investigator 49510, Lisbon
  - Site Ref # / Investigator 49513, Lisbon
  - Site Ref # / Investigator 49512, Ponta Delgada-Acores
  - Site Ref # / Investigator 26427, Ponte de Lima
- Spain (36):
  - Site Ref # / Investigator 49653, Alicante
  - Site Ref # / Investigator 49662, Asturias
  - Site Ref # / Investigator 49684, Barcelona
  - Site Ref # / Investigator 49680, Barcelona
  - Site Ref # / Investigator 49646, Barcelona
  - Site Ref # / Investigator 49645, Barcelona
  - Site Ref # / Investigator 49649, Barcelona
  - Site Ref # / Investigator 49647, Barcelona
  - Site Ref # / Investigator 49670, Barcelona
  - Site Ref # / Investigator 49667, Cadiz
  - Site Ref # / Investigator 49693, Cadiz
  - Site Ref # / Investigator 5594, Castellon
  - Site Ref # / Investigator 49663, Córdoba
  - Site Ref # / Investigator 49652, Elche
  - Site Ref # / Investigator 49651, Granada
  - Site Ref # / Investigator 49681, Granada
  - Site Ref # / Investigator 49695, Guadalajara
  - Site Ref # / Investigator 49669, Jaén
  - Site Ref # / Investigator 49689, Lleida
  - Site Ref # / Investigator 49686, Madrid
  - Site Ref # / Investigator 49697, Madrid
  - Site Ref # / Investigator 49679, Madrid
  - Site Ref # / Investigator 49650, Madrid
  - Site Ref # / Investigator 49683, Madrid
  - Site Ref # / Investigator 49687, Madrid
  - Site Ref # / Investigator 49692, Madrid
  - Site Ref # / Investigator 49664, Madrid
  - Site Ref # / Investigator 49696, Madrid
  - Site Ref # / Investigator 49665, Málaga
  - Site Ref # / Investigator 49691, Málaga
  - Site Ref # / Investigator 49685, Mostoles-Madrid
  - Site Ref # / Investigator 49666, Sant Joan Despi (Barcelona)
  - Site Ref # / Investigator 49688, Seville
  - Site Ref # / Investigator 49694, Toledo
  - Site Ref # / Investigator 49654, Valencia
  - Site Ref # / Investigator 49648, Vic (Barcelona)
- United Kingdom (6):
  - Site Ref # / Investigator 49485, Brighton
  - Site Ref # / Investigator 49470, Greater Manchester
  - Site Ref # / Investigator 49471, Harrogate
  - Site Ref # / Investigator 49476, Manchester
  - Site Ref # / Investigator 49486, Oxford
  - Site Ref # / Investigator 49472, Wigan

REFERENCES:
- [Derived] Burmester GR, Matucci-Cerinic M, Mariette X, Navarro-Blasco F, Kary S, Unnebrink K, Kupper H. Safety and effectiveness of adalimumab in patients with rheumatoid arthritis over 5 years of therapy in a phase 3b and subsequent postmarketing observational study. Arthritis Res Ther. 2014 Jan 27;16(1):R24. doi: 10.1186/ar4452. PMID 24460746

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants were treated with commercially available adalimumab in normal clinical practice.
Period: Overall Study
Arm/Group | Adalimumab
Started | 3435
Completed | 1805
Not Completed | 1630

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab
Number analyzed (Participants) | 3435
Age Continuous [Mean (Standard Deviation); unit: years] | 54.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2724
  Male | 711
Region of Enrollment [Number; unit: participants]
  Portugal | 55
  France | 689
  Greece | 232
  Spain | 476
  Belgium | 318
  Australia | 20
  Austria | 95
  Netherlands | 248
  Germany | 561
  United Kingdom | 69
  Italy | 672

OUTCOME MEASURES:

1. Primary Outcome: Disease Activity Score in 28 Joints (DAS28) Based on Erythrocyte Sedimentation Rate (ESR)
Description: DAS28 is a composite measure of disease activity in patients with rheumatoid arthritis. It is calculated on the basis of tender and swollen joint counts (each assessed in 28 joints), the patient's ESR, and the patient's subjective assessment of disease activity (assessed using a 100-mm visual analog scale). A DAS28 less than 3.2 indicates low disease activity and a DAS28 greater than 5.1 indicates high disease activity; there is no absolute range of scores due to inter-patient variability in ESR.
Time Frame: Baseline, Months 12, 24, 36, 48, and 60, and Last Observed Value
Population: Results are presented as observed. The number of participants evaluated is indicated for each time point below.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 3435
units on a scale
  Baseline of NCT00448383 (Study M02-497) (N = 3407) | 6.0 (1.1)
  Baseline of NCT00234884 (Study M03-634) (N = 2746) | 3.3 (1.3)
  Month 12 (N = 2430) | 3.1 (1.3)
  Month 24 (N = 2033) | 3.0 (1.3)
  Month 36 (N = 1746) | 3.0 (1.2)
  Month 48 (N = 1518) | 2.9 (1.2)
  Month 60 (N = 1255) | 2.8 (1.2)
  Last Observed Value (N = 3281) | 3.3 (1.5)

2. Primary Outcome: American College of Rheumatology 20% (ACR20) Response Rate
Description: ACR20 response is a 20% or better improvement from Baseline in tender joint count, swollen joint count, and at least 3 of the following 5 parameters: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire Disability Index (HAQ-DI), and C-reactive protein. Response was calculated based on values at Baseline of NCT00448383 (Study M02-497).
Time Frame: Baseline, Months 12, 24, 36, 48, and 60, and Last Observed Value
Population: Results are presented as observed. The number of participants evaluated is indicated for each time point below.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 3435
percentage of participants
  Baseline of NCT00234884 (Study M03-634) (N = 2886) | 80.3
  Month 12 (N = 2508) | 82.9
  Month 24 (N = 2116) | 84.5
  Month 36 (N = 1811) | 84.8
  Month 48 (N = 1572) | 85.8
  Month 60 (N = 1309) | 87.9
  Last Observed Value (N = 3236) | 75.8

3. Primary Outcome: American College of Rheumatology 50% (ACR50) Response Rate
Description: ACR50 response is a 50% or better improvement from Baseline in tender joint count, swollen joint count, and at least 3 of the following 5 parameters: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire Disability Index (HAQ-DI), and C-reactive protein. Response was calculated based on values at Baseline of NCT00448383 (Study M02-497).
Time Frame: Baseline, Months 12, 24, 36, 48, and 60, and Last Observed Value
Population: Results are presented as observed. The number of participants evaluated is indicated for each time point below.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 3435
percentage of participants
  Baseline of NCT00234884 (Study M03-634) (N = 2873) | 58.8
  Month 12 (N = 2509) | 62.9
  Month 24 (N = 2109) | 66.6
  Month 36 (N = 1797) | 66.2
  Month 48 (N = 1564) | 68.3
  Month 60 (N = 1293) | 70.1
  Last Observed Value (N = 3238) | 55.8

4. Primary Outcome: American College of Rheumatology 70% (ACR70) Response Rate
Description: ACR70 response is a 70% or better improvement from Baseline in tender joint count, swollen joint count, and at least 3 of the following 5 parameters: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, Health Assessment Questionnaire Disability Index (HAQ-DI), and C-reactive protein. Response was calculated based on values at Baseline of NCT00448383 (Study M02-497).
Time Frame: Baseline, Months 12, 24, 36, 48, and 60, and Last Observed Value
Population: Results are presented as observed. The number of participants evaluated is indicated for each time point below.
Measure: Number; unit: participants
Arm/Group | Adalimumab
Number analyzed (Participants) | 3435
participants
  Baseline of NCT00234884 (Study M03-634) (N = 2889) | 34.9
  Month 12 (N = 2497) | 40.2
  Month 24 (N = 2106) | 42.9
  Month 36 (N = 1786) | 44.1
  Month 48 (N = 1554) | 47.0
  Month 60 (N = 1297) | 47.5
  Last Observed Value (N = 3240) | 37.0

5. Primary Outcome: Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: HAQ-DI is a composite measure of physical function calculated on the basis of 20 questions in 8 domains (dressing, arising, eating, walking, hygiene, reach, grip, and common activities), each evaluated on a 4-point scale ranging from 0 (without any difficulty) to 3 (unable to do). HAQ-DI score is the sum of worst scores in each domain divided by the number of domains answered, and ranges from 0 (no difficulty) to 3 (unable to do). A mean change of -0.22 is considered the minimum clinically important change. Mean change in HAQ-DI was calculated from Baseline of NCT00448383 (Study M02-497).
Time Frame: Baseline, Months 12, 24, 36, 48, and 60, and Last Observed Value
Population: Results are presented as observed. The number of participants evaluated is indicated for each time point below.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab
Number analyzed (Participants) | 3435
units on a scale
  Baseline of NCT00234884 (Study M03-634) (N = 2976) | -0.70 (0.65)
  Month 12 (N = 2590) | -0.72 (0.66)
  Month 24 (N = 2177) | -0.74 (0.68)
  Month 36 (N = 1863) | -0.75 (0.68)
  Month 48 (N = 1622) | -0.76 (0.70)
  Month 60 (N = 1348) | -0.74 (0.69)
  Last Observed value (N = 3322) | -0.65 (0.73)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 5 years. For participants who discontinued the study early, investigators were asked to record adverse events up to 3 months after last dose of adalimumab.
Arm/Group | Adalimumab
Serious Adverse Events (participants affected / at risk) | 755/3435
Other Adverse Events (participants affected / at risk) | 562/3435
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Adalimumab (N=3435)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 2 (2)
Lymphoadenopathy (Blood and lymphatic system disorders) | 2 (2)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 (2)
Microcytic anaemia (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Splenic haemorrhage (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 8 (8)
Angina pectoris (Cardiac disorders) | 12 (12)
Angina unstable (Cardiac disorders) | 2 (2)
Aortic valve incompetence (Cardiac disorders) | 1 (2)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 17 (20)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 9 (11)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 9 (11)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 10 (10)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Hypertensive heart disease (Cardiac disorders) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 25 (25)
Myocardial ischaemia (Cardiac disorders) | 6 (6)
Pericardial effusion (Cardiac disorders) | 5 (5)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Tachycardia paroxysmal (Cardiac disorders) | 1 (1)
Branchial cyst (Congenital, familial and genetic disorders) | 1 (1)
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1 (1)
Odontogenic cyst (Congenital, familial and genetic disorders) | 1 (1)
Polydactyly (Congenital, familial and genetic disorders) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Cushing's syndrome (Endocrine disorders) | 1 (1)
Goitre (Endocrine disorders) | 3 (3)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 3 (3)
Cataract (Eye disorders) | 3 (3)
Entropion (Eye disorders) | 1 (1)
Macular degeneration (Eye disorders) | 1 (1)
Optic ischaemic neuropathy (Eye disorders) | 1 (1)
Retinal degeneration (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (2)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 2 (2)
Anorectal stenosis (Gastrointestinal disorders) | 1 (1)
Caecitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Colitis collagenous (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (8)
Diverticular perforation (Gastrointestinal disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Duodenal fistula (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 4 (4)
Intestinal infarction (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 4 (4)
Peritonitis (Gastrointestinal disorders) | 1 (1)
Polyp colorectal (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 4 (4)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 8 (8)
Death (General disorders) | 3 (3)
Device dislocation (General disorders) | 5 (5)
Device occlusion (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 4 (4)
Pyrexia (General disorders) | 9 (9)
Soft tissue inflammation (General disorders) | 1 (1)
Sudden death (General disorders) | 2 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
Biliary cirrhosis primary (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 7 (7)
Cholecystitis acute (Hepatobiliary disorders) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 18 (20)
Hepatic failure (Hepatobiliary disorders) | 2 (2)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1)
Amyloidosis (Immune system disorders) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1)
Secondary amyloidosis (Immune system disorders) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Abscess (Infections and infestations) | 2 (2)
Abscess neck (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 2 (3)
Appendicitis (Infections and infestations) | 3 (3)
Arthritis bacterial (Infections and infestations) | 11 (12)
Atypical mycobacterial infection (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 6 (6)
Bronchopneumonia (Infections and infestations) | 4 (4)
Bursitis infective (Infections and infestations) | 3 (3)
Cellulitis (Infections and infestations) | 7 (7)
Chronic sinusitis (Infections and infestations) | 2 (2)
Cystitis (Infections and infestations) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 5 (5)
Endocarditis staphylococcal (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Extrapulmonary tuberculosis (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 6 (6)
Gastroenteritis viral (Infections and infestations) | 1 (1)
H1N1 influenza (Infections and infestations) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1)
Hepatic echinococciasis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 5 (5)
Histoplasmosis (Infections and infestations) | 1 (3)
Infected skin ulcer (Infections and infestations) | 1 (2)
Influenza (Infections and infestations) | 2 (2)
Joint tuberculosis (Infections and infestations) | 1 (1)
Leishmaniasis (Infections and infestations) | 1 (1)
Listeria sepsis (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 4 (4)
Localised infection (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Lung abscess (Infections and infestations) | 1 (1)
Lung infections (Infections and infestations) | 9 (10)
Lyme disease (Infections and infestations) | 1 (1)
Lymphadenitis bacterial (Infections and infestations) | 1 (1)
Meningitis meningococcal (Infections and infestations) | 1 (1)
Mucocutaneous leishmaniasis (Infections and infestations) | 1 (1)
Mycobacterium avium complex infection (Infections and infestations) | 2 (2)
Mycobacterium fortuitum infection (Infections and infestations) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1)
Oseophageal candidiasis (Infections and infestations) | 1 (1)
Orchitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 3 (4)
Parainfluenzae virus infection (Infections and infestations) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1)
Peritoneal tuberculosis (Infections and infestations) | 1 (1)
Peritonsillar abscess (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pleurisy viral (Infections and infestations) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 42 (44)
Pneumonia legionella (Infections and infestations) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 3 (3)
Pseudomembranous colitis (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 3 (3)
Pyelonephritis (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 4 (4)
Pyothorax (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 7 (8)
Salmonellosis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 10 (10)
Septic arthritis staphylococcal (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Staphylococcal osteomyelitis (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 11 (11)
Urosepsis (Infections and infestations) | 3 (3)
Vaginal abscess (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Viral pericarditis (Infections and infestations) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Visceral leishmaniasis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 6 (6)
Disseminated tuberculosis (Infections and infestations) | 2 (2)
Erysipelas (Infections and infestations) | 13 (15)
Escherichia sepsis (Infections and infestations) | 2 (2)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 5 (5)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2)
Decompression sickness (Injury, poisoning and procedural complications) | 1 (1)
Diffuse axonal injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 9 (9)
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 (6)
Femur fracture (Injury, poisoning and procedural complications) | 7 (7)
Fibula fracture (Injury, poisoning and procedural complications) | 3 (3)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4)
Foreign body (Injury, poisoning and procedural complications) | 1 (1)
Fractured ischium (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 2 (2)
Graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 9 (9)
Humerus fracture (Injury, poisoning and procedural complications) | 6 (7)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 (4)
Meniscus lesion (Injury, poisoning and procedural complications) | 2 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 2 (2)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 2 (2)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2)
Splenic injury (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 2 (2)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 6 (6)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 3 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 4 (4)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Antiphospholipid antibodies (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood amylase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 2 (2)
Mycobacterium test positive (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Central obesity (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Bone formation decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Felty's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 8 (8)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 5 (5)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint destruction (Musculoskeletal and connective tissue disorders) | 4 (4)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 (19)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pseudarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 7 (7)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (6)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 3 (3)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
B-cell lymphoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellopontine angle tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Conjunctival melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glomus jugulare tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian granulosa-theca cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Primary mediastinal large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (10)
Amnestic disorder (Nervous system disorders) | 1 (1)
Amyotrophic lateral sclerosis (Nervous system disorders) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 2 (2)
Cerebellar atrophy (Nervous system disorders) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 4 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 11 (11)
Cervical myelopathy (Nervous system disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1)
Coma (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Facial palsy (Nervous system disorders) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Hypoglycaemic coma (Nervous system disorders) | 1 (1)
Hypoxic encephalopathy (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 5 (5)
Loss off consciousness (Nervous system disorders) | 2 (2)
Mononeuropathy multiplex (Nervous system disorders) | 1 (1)
Optic neuritis (Nervous system disorders) | 2 (2)
Parkinson's disease (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 4 (4)
Speech disorder (Nervous system disorders) | 1 (1)
Transient global amnesia (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 6 (6)
Vascular dementia (Nervous system disorders) | 1 (1)
Vascular encephalopathy (Nervous system disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Placenta previa (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 4 (5)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 5 (6)
Calculus urinary (Renal and urinary disorders) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 3 (3)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 7 (7)
Renal failure acute (Renal and urinary disorders) | 7 (7)
Ureteric rupture (Renal and urinary disorders) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 1 (2)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Breast cyst (Reproductive system and breast disorders) | 1 (1)
Breast enlargement (Reproductive system and breast disorders) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2)
Cystocele (Reproductive system and breast disorders) | 3 (3)
Genital prolapse (Reproductive system and breast disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Pelvic fluid collection (Reproductive system and breast disorders) | 1 (1)
Prostatic disorder (Reproductive system and breast disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 3 (3)
Rectocele (Reproductive system and breast disorders) | 2 (2)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 5 (5)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Anoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal tubinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia effluvium (Skin and subcutaneous tissue disorders) | 1 (1)
Cutaneous lupus erythematosis (Skin and subcutaneous tissue disorders) | 2 (2)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1)
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 3 (3)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 5 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1)
Blepharoplasty (Surgical and medical procedures) | 1 (1)
Removal of internal fixation (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 2 (2)
Aortic stenosis (Vascular disorders) | 2 (2)
Arterial haemorrhage (Vascular disorders) | 2 (2)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Arteritis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 5 (5)
Haematoma (Vascular disorders) | 1 (1)
Haemodynamic instability (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypertensive crisis (Vascular disorders) | 3 (4)
Hypotension (Vascular disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (3)
Phlebitis (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (4)
Varicose vein (Vascular disorders) | 1 (1)
Vasculitis (Vascular disorders) | 2 (2)
Venous insufficiency (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab (N=3435)
Bronchitis (Infections and infestations) | 244
Nasopharyngitis (Infections and infestations) | 189
Urinary tract infection (Infections and infestations) | 195

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.